CLINICAL TRIAL: NCT07247799
Title: Ozone Therapy for the Treatment of Oral Mucositis in Patients Undergoing Radio and Chemotherapy in the Head and Neck Region: Retrospective Observational Study
Brief Title: Ozone Therapy for the Treatment of Oral Mucositis in Patients Undergoing Radio and Chemotherapy in the Head and Neck Region
Status: Completed | Type: Observational
Sponsor: Andrea Scribante (Other)
Responsible Party: Sponsor-Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Organization: University of Pavia (Other)
Other Study IDs: 2025-OZONEMUCOSITIS
Record Dates: First submitted 2025-11-14; First posted 2025-11-25 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Oral Mucositis; Head and Neck Neoplasms
MeSH Terms: conditions — Stomatitis; Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients undergoing radio and chemotherapy for head and neck cancer
  Interventions: Device: Ozone treatment
- Patients undergoing radio and chemotherapy for cancers in other districts
  Interventions: Device: Ozone treatment

INTERVENTIONS:
Device: Ozone treatment — Ozone DTA (Sweden & Martina SpA, 35020 Due Carrare, PD, Italy) for clinical application; home oral care with DentO3® toothpaste, CollutO3®, Ozoral® Gel (Innovares, Sant'Ilario d'Enza (RE) - Italy).

SUMMARY:
The present study aims to evaluate the effectiveness of a combined protocol of professional and at-home ozone therapy in the treatment of oral mucositis in patients undergoing radio- and/or chemotherapy.

In-office treatment was performed using a medical ozone generator, while at-home therapy involved the daily application of high-concentration ozonated oil products. The study assessed the reduction in mucositis severity (WHO scale), decrease in pain (VAS scale), and improvement in patient-reported quality of life, with specific attention to nutrition, oral hygiene, and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing radio and chemotherapy for head and neck cancer and cancers in other districts

Exclusion Criteria:

* syndromic patients
* pregnant women
* patients with cardiac pacemakers
* epileptic patients
* patients with high sensitivity to electric current

Ages: 40 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients under orthodontic care at the Section of Dentistry
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
WHO scale for oral mucositis | At baseline (T0), baseline after treatment (T1), after 48 hours (T2), at day five (T3), at day eight (T4), at day twelve (T5), at day fifteen (T6)
  Scoring criteria:
  * 0 None
  * 1 Oral soreness, erythema
  * 2 Oral erythema, ulcers, solid diet tolerated
  * 3 Oral ulcers, liquid diet only

SECONDARY OUTCOMES:
Visual Analogue Scale | At baseline (T0), baseline after treatment (T1), after 48 hours (T2), at day five (T3), at day eight (T4), at day twelve (T5), at day fifteen (T6)
  Evaluation of self-perceived pain from 0 (no pain) to 10 (worst pain ever)
Questionnaire | At baseline (T0) and at day fifteen (T6)
  Score from 0=best outcome to 10= worst outcome for the following items:
  * On a scale from 1 to 10, how much discomfort do certain foods and beverages cause you?
  * On a scale from 1 to 10, to what extent does your oral condition make you limit the intake of certain foods and beverages?
  * On a scale from 1 to 10, how much do certain food textures (e.g., crunchy foods) bother you?
  * On a scale from 1 to 10, to what extent does your oral condition lead you to limit the texture of the foods you consume?
  * On a scale from 1 to 10, how much discomfort does the temperature of certain foods and beverages cause you?
  * On a scale from 1 to 10, to what extent does your oral condition make you limit the temperature of the foods and beverages you consume?
  * On a scale from 1 to 10, how much does your oral condition cause discomfort during your daily oral activities?
  * On a scale from 1 to 10, how much discomfort does your oral condition cause during daily oral hygiene (brushin

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy